CLINICAL TRIAL: NCT06820619
Title: Efficacy of Mindfulness-based Training for Teachers and Young Children for Social Emotional and Ethical Development (SEED)-Randomized Controlled Trial
Brief Title: Efficacy of Mindfulness-based Training for Teachers and Young Children for Social Emotional and Ethical Development (SEED)
Acronym: SEED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Xi'an Jiaotong-Liverpool University (Unknown)
Responsible Party: Principal Investigator, Winnie W.S. MAK, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SBRE-22-0785B
Record Dates: First submitted 2024-11-29; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-11

CONDITIONS: Development, Child; Mindfulness; Wellbeing
Keywords: social, emotional, and ethical development; mindfulness; mental well-being; young children
MeSH Terms: conditions — Psychological Well-Being | interventions — Seeds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Social, Emotional, and Ethical Development (SEED) curriculum (Experimental): The kindergarten teachers and children will receive training and 12-week SEED curriculum. Upon informed consent from the school principals and parents, teachers will receive mindfulness training and complete pre- and post-training assessments, and a one-month follow-up assessments. Teachers will be taught 8 mindfulness exercise to integrate into the daily teaching and students in intervention group will receive a 30-min lesson of SEED curriculum per week, 12-weeks in total, lead by the Bohdi Love Foudation tutors. Parents and students will complete questionnaries and assessments pre- and post-intervention.
  Interventions: Behavioral: Social, Emotional, and Ethical Development (SEED) curriculum
- Waitlist control group (No Intervention): Two kindergartens will be assigned to the waitlist control condition. Teachers in the waitlist control schools will wait for at least 12 weeks before they receive the training, and children in the waitlist control group will receive SEED curriculum after the teachers' training. Upon informed consent from the school principals and parents, teachers will complete pre-, post-, and 4-week follow-up assessments about their mindfulness and relevant concept. Parents will complete pre- and post- questionnaires about the adjustment of the child. Children will complete pre- and post- assessment tasks with experimenters.

INTERVENTIONS:
Behavioral: Social, Emotional, and Ethical Development (SEED) curriculum — In response to fulfilling children's urgent psychosocial needs, the Bodhi Love Foundation (BLF) adapted the Kindness Curriculum for young children in Hong Kong by translating it from English to Chinese and adapting its length and content for implementation in the local kindergarten context. The adapted Kindness Curriculum, renamed as Social, Emotional, and Ethical Development curriculum (SEED), is a two-part program involving teacher training and delivery of SEED. The teacher training is consist of a 12-hour mindfulness course and a 1-day (6 hours) workshop to get familiarized with the understanding and practice of mindfulness, and the details of the SEED Curriculum. The SEED Curriculum involves 8 short sessions of basic techniques in mindfulness with 10 minutes each. In addition, it has 12 mindfulness-based lessons with specific themes for children in K1 and K2. Each lesson lasts for approximately 30-40 minutes.
  Arms: Social, Emotional, and Ethical Development (SEED) curriculum

SUMMARY:
The objectives of the present study are to (1) evaluate the effectiveness of implementing teachers' training on mindfulness and developing their competency in delivering the Social, Emotional, and Ethical Development (SEED) curriculum to preschool children and (2) evaluate the effectiveness of the SEED curriculum at kindergartens in improving children's well-being and related outcomes. Randomized controlled trials will be conducted to investigate the effectiveness of SEED teacher training and the SEED Curriculum. A minimum of four kindergartens will be recruited to participate in the study. Half of the kindergartens, teachers, and children will receive the training and SEED curriculum, while the other half will be assigned to the waitlist control condition. Upon informed consent from the school principals and parents, teachers will receive mindfulness training and complete pre- and post-training assessments, and one-month follow-up assessments. Teachers will be taught 8 mindfulness exercises to be integrated into daily teaching and students in the intervention group will receive a 30-minute lesson of SEED curriculum per week, 12 weeks in duration, led by the Bodhi Love Foundation SEED trainers. Parents and students will complete assessments before intervention and after intervention(in the 12th week).

DETAILED DESCRIPTION:
According to the World Health Organization, early child development lays a critical foundation for healthy habits and long-term development, including health and well-being, as well as changing the trajectory of the next generation in maximizing human potential. Specifically, social-emotional learning (SEL) in early childhood lays the foundation for their later adjustment, including better emotional wellness and fewer internalizing and externalizing problems. Recently, numerous SEL programs have been developed worldwide. Among these evidence-based SEL programs, the Kindness Curriculum is a secular mindfulness-based SEL program designed for children between 4-6 years of age.

In Hong Kong, the Kindergarten Education Curriculum Guide has identified affective and social development as a major objective in early childhood. Better social-emotional competence is associated with preschool-aged children's lower anxiety and fewer aggressive behaviors in Hong Kong. However, the implementation of evidence-based SEL programs remains immature, with very few programs available for kindergartens and kindergarten-cum-child care settings and none being mindfulness-based. In response to fulfilling children's psychosocial needs, the Bodhi Love Foundation (BLF) has adapted the Kindness Curriculum for young children in Hong Kong. With the concerted efforts of a team of qualified local mindfulness teachers and Prof. Daniel Goleman as the advisor, the curriculum was translated from English to Chinese and has been adapted for implementation in the local cultural context. The adapted Kindness Curriculum, renamed as Social, Emotional, Ethical Development Curriculum (SEED), is a two-part program involving training teachers on mindfulness and delivery of SEED to young children. As such, the curriculum may be beneficial for both teachers and children.

The project's significance is to cultivate mindfulness and loving-kindness among our teachers and children to equip them with the mindset and skills needed for self-care and the promotion of mental well-being. Such well-being promotion and distress prevention approach that starts early in childhood lays a critical cornerstone for children to develop healthily, which can potentially reduce the incidence of mental illness among younger generations.

ELIGIBILITY:
Inclusion Criteria:

* For children: aged 3-7 years old, understand Cantonese
* For parents: aged 18 years old or above, understand Cantonese
* For teachers: aged 18 years old or above, understand Cantonese, currently working at a kindergarten

Exclusion Criteria:

* Cannot understand Cantonese

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mindfulness in Teaching Scale(MTS) | Pre-intervention assessment, Post-intervention assessment at 6th week, follow up assessment at 10th week
  The 14-item Mindfulness in Teaching Scale(MTS) will be used to assess the extent to which teachers are consciously aware of various classroom and student activities. It contains 2 subscales measuring teacher intrapersonal and interpersonal mindfulness. Items are answered on a 5-point Likert scale (from 1 = never, to 5 = always). The total score of each dimension is obtained by summing the respective items, with higher scores indicating greater levels of Teacher Intrapersonal Mindfulness (ranging from 9 to 45) and Teacher Interpersonal Mindfulness (ranging from 5 to 25).
Copenhagen Burnout Inventory | Pre-intervention assessment, Post-intervention assessment at 6th week, follow up assessment at 10th week
  he personal burnout and work-related burnout subscale in Copenhagen Burnout Inventory (CBI) will be used to measure teachers' burnout in three domains: and client-related burnout. CBI shows good reliability for each subscale (Cronbach's alpha = .85-.87).
The Impermanence Awareness and Acceptance Scale | Pre-intervention assessment, Post-intervention assessment at 6th week, follow up assessment at 10th week
  The 13-item Impermanence Awareness and Acceptance Scale (IMAAS) measures changes in an individual's state levels of impermanence awareness and impermanence acceptance on a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree).
Interconnectedness Scale | Pre-intervention assessment, Post-intervention assessment at 6th week, follow up assessment at 10th week
  The 12-item Interconnectedness Scale will be used to measure participants' awareness on their interdependent relationship with all matters in the world on a 6-point scale from 1 (totally disagree) to 6 (totally agree). The scale measures interconnectedness in three dimensions: emotional response to interconnectedness, appreciation of interconnectedness on self-development, and interconnectedness in social relations.
Mindfulness-Discernment Scale (MDS) | Pre-intervention assessment, Post-intervention assessment at 6th week, follow up assessment at 10th week
  The 20-item Five Facet Mindfulness Questionnaire Short Form (FFMQ-SF) and 10-item Mindfulness subscale in the Mindfulness-Discernment Scale will be used to measure levels of mindfulness. FFMQ-SF measures five dimensions of mindfulness including observing, describing, acting with awareness, nonjudging, and nonreactivity (Baer et al., 2008) on a 5-point Likert scale ranging from 1 (never) to 5 (always). Discernment will be assessed using the 14-item Discernment subscale in the Mindfulness-Discernment Scale. Items are rated on a scale ranging from 1 (Never) to 6 (Always).
Nonattachment Scale(NAS)-Short Form | Pre-intervention assessment, Post-intervention assessment at 6th week, follow up assessment at 10th week
  The 8-item Nonattachment Scale Short Form will be used to assess participants' flexibility and balanced approach towards life experiences on a 6-point scale. Participants rated the items from 1 (disagree strongly) to 6 (agree strongly). Three items were reversed-coded and higher scores indicate higher level of nonattachment. This abridged version was developed and validated using item response theory in Hong Kong Chinese sample.
Santa Clara Brief Compassion Scale | Pre-intervention assessment, Post-intervention assessment at 6th week, follow up assessment at 10th week
  The Santa Clara Brief Compassion Scale (SCBCS) is a 5-item inventory that measures compassion for others using a 7-point Likert-like scale (1 = not at all true of me to 7= very true of me), which yields a possible range of 5 to 35 points, with higher scores mean a higher level of compassion.
The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) | Pre-intervention assessment, Post-intervention assessment at 6th week, follow up assessment at 10th week
  Warwick-Edinburgh Mental Wellbeing Scale-Short is a 7-item self-report measure of subjective mental well-being on a 5-point Likert scale (1=none of the time, 5=all of the time), giving a minimum score of 14 and maximum score of 70. A higher WEMWBS score therefore indicates a higher level of mental well-being. The Chinese translation has demonstrated high levels of internal consistency, test-retest reliability, and construct validity in both community and clinical samples.
Strengths and Difficulties Questionnaire (SDQ) | Pre-intervention assessment, Post-intervention assessment at 12th week
  A 20-item internalizing and externalizing problems subscales of the Strengths and Difficulties Questionnaire will be used to access their child's adjustment difficulties on a 3-point scale ranging from 1 (not true) to 3 (certainly true). The internalizing problems subscale capture emotional symptoms and peer relationship problems, whereas the externalizing problems subscale capture conduct problems and hyperactivity/inattention.
Social Skills Improvement System-Rating Scales (Preschool Parents version) (SSIS - SEL) | Pre-intervention assessment, Post-intervention assessment at 12th week
  The SSIS SEL consists of 20 items which assess children's skills in each of the five social-emotional learning competencies: Self-Awareness, Self-Management, Social Awareness, Relationship Skills, Responsible Decision Making.
Child Prosocial Behavior Questionnaire (CPBQ) | Pre-intervention assessment, Post-intervention assessment at 12th week
  CPBQ consists of 10 items, Parents are asked to rate their child on a 5-point likert scale ranging from 1(never) to 5(always) on prosocial behaviors. CPBQ consists 3 subscales, 1.Sharing, examples include:"Willingly shares toys with a parent, even without being asked". 2. Comforting, examples include: "Hugs others when they are upset". 3.Helping:"Picks up something that I have accidentally dropped and hands it to me"
Children's Behavioral Questionnaire(CBQ) age 3-7-Short Form | Pre-intervention assessment, Post-intervention assessment at 12th week
  In the CBQ, parents are asked to rate their child on a 7-point scale ranging from 1 (extremely untrue of your child) to 7 (extremely true of your child). Parents are also provided with a Not Applicable response option when the child has not been observed in the situation described. The standard form consists 15 subscales, in this study, 3 subscales (18 items in total) from short form are used, namely Attentional Control, Impulsivity, and Inhibitory Control. A higher score on each subscale reflects a greater level of attentional control, Impulsivity, and Inhibitory Control, respectively.
Delay of Shared Gratification Task | Pre-intervention assessment, Post-intervention assessment at 12th week
  The 5-minute Delay of Shared Gratification Task measures children's sharing behavior involving the small stickers. Children will be asked to share 1-2 stickers with other people over four instances, such as sharing with cost, sharing without cost, and delay of sharing.
Dictator game experiment | Pre-intervention assessment, Post-intervention assessment at 12th week
  Children are given 10 stickers and told these 10 belong to them. Then they were told that the other child would come in that day but would not get stickers. Children then chose how many of their stickers to share with an anonymous other child (gender matched). To give children privacy, the experimenter then closed his or her eyes while children put the stickers they wanted to keep in their envelope and put the stickers they wanted to give away in the envelope for the other child. Experimenter count the number of stickers that's given to the "other child".
Puppet Task | Pre-intervention assessment, Post-intervention assessment at 12th week
  Children will play 3 games alongside a puppet. In each game the puppet/adult realized that they did not have sufficient pieces to finish the task and became distressed that they were unable to receive a sticker. There were three distress prompts, which increased in the emotional intensity of suffering shown, This allowed three opportunities for the child to help. Helping was coded per task on a scale of 0(didn't help)-4(helped with no prompting). The total helping score could get is 0-12. if the child did not help, whether they console or disengage with the puppet is also coded.

CONTACTS AND LOCATIONS:
Overall Officials: Winnie WS MAK, Principal Investigator — Chinese University of Hong Kong; Rebecca YM Cheung, Principal Investigator — Xi'an Jiaotong-Liverpool University
Locations (1):
- Dept of Psychology, CUHK, Hong Kong,, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blewitt C, Fuller-Tyszkiewicz M, Nolan A, Bergmeier H, Vicary D, Huang T, McCabe P, McKay T, Skouteris H. Social and Emotional Learning Associated With Universal Curriculum-Based Interventions in Early Childhood Education and Care Centers: A Systematic Review and Meta-analysis. JAMA Netw Open. 2018 Dec 7;1(8):e185727. doi: 10.1001/jamanetworkopen.2018.5727. PMID 30646283
- [Background] Green M, Kirby JN, Nielsen M. The cost of helping: An exploration of compassionate responding in children. Br J Dev Psychol. 2018 Nov;36(4):673-678. doi: 10.1111/bjdp.12252. Epub 2018 Jun 10. PMID 29888498
- [Background] Flook L, Goldberg SB, Pinger L, Bonus K, Davidson RJ. Mindfulness for teachers: A pilot study to assess effects on stress, burnout and teaching efficacy. Mind Brain Educ. 2013 Sep;7(3):10.1111/mbe.12026. doi: 10.1111/mbe.12026. PMID 24324528
- [Background] Dunning D, Tudor K, Radley L, Dalrymple N, Funk J, Vainre M, Ford T, Montero-Marin J, Kuyken W, Dalgleish T. Do mindfulness-based programmes improve the cognitive skills, behaviour and mental health of children and adolescents? An updated meta-analysis of randomised controlled trials. Evid Based Ment Health. 2022 Jul 12;25(3):135-42. doi: 10.1136/ebmental-2022-300464. Online ahead of print. PMID 35820989